CLINICAL TRIAL: NCT07323823
Title: The Effect of 850 nm Photobiomodulation Therapy (PBM) on the Electrical Activity of the Brain in Stroke Patients
Brief Title: The Effect of PBM on the Electrical Activity of the Brain in Stroke Patients
Acronym: PBM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Yong-il Shin, PhD, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-2025-009
Record Dates: First submitted 2025-12-22; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Post-stroke Aphasia
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Experimental Group (850nm PBM + Standard Rehabilitation) (Experimental)
  Interventions: Device: photobiomodulation (PBM); Other: control group-receive speech therapy
- Arm 2: Control Group ( Standard Rehabilitation) (Sham Comparator)
  Interventions: Other: control group-receive speech therapy

INTERVENTIONS:
Device: photobiomodulation (PBM) — Experimental Group: Participants will receive iSyncWave transcranial photobiomodulation (tPBM) and speech therapy, with 20 minutes per modality per session, once daily, 5 days per week, for 4 weeks, totaling 20 sessions of combined intervention. During the intervention period, changes in concomitant medications and concurrent therapies will be monitored and recorded; any modifications to medications or therapies must be documented in detail.
  Arms: Arm 1: Experimental Group (850nm PBM + Standard Rehabilitation)
Other: control group-receive speech therapy — Participants will receive speech therapy at a frequency of 20 minutes per session, once daily, 5 days per week, for 4 weeks, with a total of 20 sessions.

SUMMARY:
The Effect of Low-Level Light Therapy on the Electrical Activity of the Brain in Stroke Patients

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with ischemic or hemorrhagic stroke by a specialist. Patients in the recovery phase within 1 year after onset; those with confirmed clinical functional impairment upon assessment, who are conscious and able to cooperate with PBM stimulation and evaluations.

Adult patients (≥ 18 years old) ，less than 80 years old，who have signed the informed consent form, or patients with proxy consent.

Exclusion Criteria:

* Individuals with photosensitive skin at risk of developing urticaria or dermatitis.

Patients judged to have an unstable surgical site following hemorrhagic stroke-related surgery.

Pregnant or lactating individuals. Individuals with a history of seizures. Individuals who have participated in clinical studies twice or more in the same year or in other clinical studies within 6 months.

Other individuals with clinically significant findings deemed medically inappropriate for the study by the principal investigator or responsible researcher.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
electroencephalography (EEG) | Change in from baseline to post 20 sessions (up to approximately 4 weeks) α-Wave Increased amplitude, β-Wave moderate amplitude enhancement and θ-Wave Decreased excessive amplitude indicate functional recovery.

SECONDARY OUTCOMES:
Korean-Western Aphasia Battery(K-WAB) | Change in Korean-Western Aphasia Battery from baseline to post 20 sessions (up to approximately 4 weeks), Higher scores indicate better language function(Total score range: 0-100 points).
Boston Naming Test (BNT) | Change in Boston Naming Test from baseline to post 20 sessions (up to approximately 4 weeks), Higher scores indicate better naming ability(Total score range: 0-60 points).
K-MMSE (Korean-Mini-Mental State Examination) | Change in K-MMSE (Korean-Mini-Mental State Examination) from baseline to post 20 sessions (up to approximately 4 weeks), Higher scores indicate better global cognitive function(Total score range: 0-30 points).
K-MoCA (Korean-Montreal Cognitive Assessment) | Change in K-MoCA (Korean-Montreal Cognitive Assessment) from baseline to post 20 sessions (up to approximately 4 weeks), Higher scores indicate better cognitive function(Total score range: 0-30 points).
CDR ( Clinical Dementia Rating Scale) | Change in CDR ( Clinical Dementia Rating Scale) from baseline to post 20 sessions (up to approximately 4 weeks), Lower scores indicate better cognitive function(Total score range: 0-18 points).
Beck Depression Inventory | Change in Beck Depression Inventory from baseline to post 20 sessions (up to approximately 4 weeks), Lower scores indicate milder depression (The total score range is 0-63 points).
EuroQol 5-Dimension Questionnaire(EQ-5D) | Change in EuroQol 5-Dimension Questionnaire(EQ-5D) from baseline to post 20 sessions (up to approximately 4 weeks), Higher scores indicate better quality of life(Total score range: -0.171 ~ 1.000 points).

IPD SHARING:
Plan to Share IPD: Yes